CLINICAL TRIAL: NCT03765086
Title: Karydakis Procedure Vs Limberg Flap in Treatment of Sacrococcygeal Pilonidal Sinus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Medical Officer, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s7
Record Dates: First submitted 2018-07-11; First posted 2018-12-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Karydakis procedure (Active Comparator): Karydakis Procedure: In this procedure the pilonidal sinus will be excised by semilunar incision so that the incision line closure will be away from midline.
  Interventions: Procedure: Karydakis procedure
- Limberg Flap (Active Comparator): Limberg Flap: In this procedure the pilonidal sinus will be excised by diamond shaped incision and the defect will be closed by random pattern flap.
  Interventions: Procedure: Limberg Flap

INTERVENTIONS:
Procedure: Karydakis procedure — Pilonidal sinus will be excised by Karydakis procedure
  Arms: Karydakis procedure
Procedure: Limberg Flap — Pilonidal sinus will be excised by Limberg Flap
  Arms: Limberg Flap

SUMMARY:
This study will be a randomized controlled trial in which there will be comparison of the effectiveness of Karydakis procedure and Limberg flap in treatment of sacrococcygeal pilonidal sinus

ELIGIBILITY:
Inclusion Criteria:

* Patients with pilonidal sinus of any sex and aged 20 years or above
* Non infected pilonidal sinus

Exclusion Criteria:

* Infected pilonidal sinus
* Uncontrolled diabetes
* Patient on immunosuppressive therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients presenting with recurrence of pilonidal sinus | 8 to 12 weeks
  Recurrence of Pilonidal Sinus(described as appearance of multiple discharging sinuses in operative site) after surgical procedure

SECONDARY OUTCOMES:
Number of weeks in which the operative wound will be healed | 4 to 6 weeks
  Duration of wound healing (complete epithelization of wound )
percentage of patients developing postoperative pain | 3 days
  postoperative pain( measured by visual analog score with 1 being minimum score and 10 being maximum score) after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mahmmood Ayyaz, mbbs, fcps, Study Director — Services Hospital, Lahore
Locations (1):
- Services hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided